CLINICAL TRIAL: NCT06391099
Title: Phase I Study of the Safety and Feasibility of a Ketogenic Dietary Intervention to Improve Response to Immunotherapy
Brief Title: Ketogenic Dietary Intervention to Improve Response to Immunotherapy in Patients With Metastatic Melanoma and Metastatic Kidney Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Marium Husain, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-21335; NCI-2024-01894 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Cutaneous Melanoma; Metastatic Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Diet Therapy; Glucose; Ketones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Ketogenic diet) (Experimental): Patients undergo a ketogenic dietary intervention with personalized coaching from a dietician about the KD, which includes extensive educational and ongoing support on the KD and continuous ketone monitoring by talking to a dietician directly, with the ability to text a dietician at any time and expect a response within 12 hours over 24weeks. Patients also undergo daily blood glucose and ketone monitoring, undergo CT, undergo blood sample collection and may undergo stool sample collection on the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Dietary Intervention; Other: Educational Activity; Other: Glucose Measurement; Other: Ketone Measurement; Other: Questionnaire Administration
- Arm II (usual caare) (Active Comparator): Patients follow a standard of care diet on the study.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Undergo standard of care diet
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual caare)
Procedure: Biospecimen Collection — Undergo blood and stool sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm I (Ketogenic diet)
Procedure: Computed Tomography — Under CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
  Arms: Arm I (Ketogenic diet)
Other: Dietary Intervention — Undergo ketogenic diet
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm I (Ketogenic diet)
Other: Educational Activity — Receive coaching support
  Arms: Arm I (Ketogenic diet)
Other: Glucose Measurement — Undergo blood glucose testing
  Other Names: GLUC; Glucose
  Arms: Arm I (Ketogenic diet)
Other: Ketone Measurement — Undergo ketone measurement
  Other Names: Ketones
  Arms: Arm I (Ketogenic diet)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm I (Ketogenic diet)

SUMMARY:
This phase I trial studies how well a ketogenic dietary intervention works to improve response to immunotherapy in patients with melanoma and kidney cancer that has spread from where it first started (primary site) to other places in the body (metastatic). A ketogenic diet (KD) means eating fewer carbohydrates and more fats. The purpose is to use ketones (normal breakdown from fat) instead of glucose (sugar) as an energy source. Researchers want to see whether a ketogenic diet can improve tumor response in patients receiving immune checkpoint inhibitors (ICI). ICI are newer treatment options that help the immune system better fight some cancers. Following a KD may improve tumor response in patients with metastatic melanoma and metastatic kidney cancer treated with ICI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and feasibility of establishing a ketogenic dietary intervention trial with longitudinal biospecimen collection in the Ohio State University Comprehensive Cancer Center (OSUCCC) cutaneous and genitourinary oncology clinics.

EXPLORATORY OBJECTIVE:

I. To assess whether the microbiome (binary, high versus [vs] low diversity) mediates the relationship between time in ketosis (days with peripheral blood beta-hydroxybutyric acid [BHB] > 0.5 mM) and tumor size over the course of treatment.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo a ketogenic dietary intervention with personalized coaching from a dietician about the KD, which includes extensive educational and ongoing support on the KD and continuous ketone monitoring by talking to a dietician directly, with the ability to text a dietician at any time and expect a response within 12 hours over 24weeks. Patients also undergo daily blood glucose and ketone monitoring, undergo computed tomography (CT), undergo blood sample collection and may undergo stool sample collection on the study.

ARM II: Patients follow a standard of care diet on the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age >= 18 years
* Clinical site A will include patients with confirmed diagnosis of metastatic melanoma (including those with brain metastases) receiving first line treatment with combination nivolumab and ipilimumab or single agent ipilimumab, nivolumab, pembrolizumab
* Clinical site B will include patients with confirmed diagnosis of metastatic renal cell carcinoma (RCC) (including those with brain metastases) receiving first line treatment with combination nivolumab and ipilimumab or single agent PD-1 inhibitor (e.g., nivolumab, pembrolizumab)
* Scheduled for imaging every 6 to 12 weeks for metastatic melanoma (MM) and mRCC as is standard of care per National Comprehensive Cancer Network (NCCN) guidelines
* Able to read, understand, and provide written informed consent
* Willing to provide stool specimen for research studies as outlined in the timeline
* Willing to participate in a ketogenic diet (KD)

Exclusion Criteria:

* Individuals < 18 years of age
* Unable or unwilling to provide consent
* Patients with type 1 diabetes mellitus or type 2 diabetes using insulin
* Patients who are clinically underweight (body mass index [BMI] < 18.5) at the start of treatment
* Other active malignancy (other than adequately treated and cured basal or squamous cell skin cancer, curatively treated in situ disease, or any other cancer from which the patient has been disease free >=5 years)
* Currently consuming a low-carbohydrate (< 130 g/day) or ketogenic diet or done so in the last 6-months
* Women who are known to be pregnant are excluded. However no additional pregnancy testing out of what would be recommended prior to initiating anti-cancer therapy will be performed solely for this study
* Patients currently participating in an interventional or therapeutic clinical trial involving the use of active anti-cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 year
  Will be assessed by immune-related adverse events (irAEs), serious adverse events (SAEs), Treatment Emergent Adverse Events (TEAEs), clinical laboratory, vital signs, physical examinations. Will be monitored during study visits and telephone calls using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, which also includes irAEs. Grade 3, 4 and 5 toxicities will be reported as adverse events.
Adherence (feasibility measure) | Up to 1 year
  Adherence will be defined as > 80% of days in ketosis and compliant as collecting all gut microbiome specimens. Diet adherence and progress will be assessed daily using at-home whole capillary blood glucose and continuous ketone monitoring devices

CONTACTS AND LOCATIONS:
Overall Officials: Marium Husain, MD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu